CLINICAL TRIAL: NCT04013607
Title: The Study of Fiber Fermentation, and Short Chain Fatty Acid Kinetics and Utilization Inside the Gut and Systemic Circulation
Brief Title: Fiber Fermentation Kinetics Inside the Gut, and Utilization of Bacterial Metabolites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL69449.081.19
Record Dates: First submitted 2019-04-23; First posted 2019-07-10 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Metabolism; Dietary Fiber; Intestine
Keywords: short chain fatty acid; dietary fiber

STUDY DESIGN:
Intervention Model Description: All subjects will consume a NDC bolus. When fermentation has started, isotopically 13C-labelled SCFAs will be delivered inside the intestine. Thereafter, production and inter-conversion of SCFAs and breakdown of fiber will be studied in luminal samples. Also blood samples will be taken to study integration of the 13C-label into various metabolic compounds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fiber drink (Experimental): A drink high in fructo- and galacto-oligosaccharides.
  Interventions: Dietary Supplement: fructo- and galacto-oligosaccharides

INTERVENTIONS:
Dietary Supplement: fructo- and galacto-oligosaccharides — A NDC drink rich in fructo- and galacto-oligosaccharides

SUMMARY:
In this study, the life course of SCFA and their regulatory role in human metabolism will be traced using a nose-intestine catheter. The investigators have methodological questions: investigate the envisioned kinetic profiles of stable isotope tracers of SCFAs, and to establish the time points of plasma sampling (to determine systemic availability of SCFAs). The resulting timepoints established in this pilot study will be applied during a future human intervention study.

DETAILED DESCRIPTION:
Background: Nowadays there is a strong interest in optimising human health through manipulation of non-digestible carbohydrates (NDC). NDC are fermented by the microbiota, hereby producing fermentation end products, mainly short chain fatty acids (SCFA) acetate, butyrate, and propionate. It is hypothesized that SCFAs mediate parts of the beneficial effects of NDC. In mice, the influx of SCFA into the host correlated strongly with improvements of markers of the metabolic syndrome, whereas concentrations of SCFA in the cecum did not. The production and influx/incorporation of SCFAs in humans will be investigated.

Study design: At day 1 the catheter will be placed. After an overnight fast at day 2, 5 subjects will consume a NDC bolus. Isotopically 13C-labelled SCFAs will be delivered in the cecum. Samples will be taken in the cecum and blood before, and continuously after dispensing the 13C-labelled SCFAs.

Study population: 5 healthy male volunteers (18-60yrs, and BMI between 18.5-30 kg/m2).

Main study parameters/endpoints: (isotopic) enrichments of SCFAs in cecum, and label incorporation in plasma metabolites such as organic acids, glucose, cholesterol, fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age 18-60yrs
* BMI between 18.5 and 30 kg/m2
* Regular bowel movement (defaecation on average once a day)
* Signed informed consent

Exclusion Criteria:

* Having a history of medical or surgical events that, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results of the study (e.g. diabetes, cardiovascular disease, gastrointestinal disease, renal failure, cancer, infectious disease, nose/throat).
* Use of any prescribed or non-prescribed medication (other than paracetamol) including antacids, analgesics, and herbal remedies during the three (3) weeks prior to study start.
* Carrying a pacemaker or any other (implanted) medical electronic device
* Smoker
* Unstable body weight (weight gain or loss >5kg in the past 3 months prior to the study start)
* Use of antibiotics within 3 months of starting the study or planned during the study
* Use of pro- or prebiotics (e.g. galacto-oligosaccharides, fructo-oligosaccharides)
* Constipation/infrequent bowel movement
* Abuse of drugs/alcohol (alcohol: >4 consumptions/day or >21 consumptions/week)
* Participation in another biomedical study
* Having diarrhoea within 2 months prior to the study start
* Personnel of Wageningen University, Division of Human Nutrition, their partner and their first and second degree relatives
* Current participation in other research from the Division of Human Nutrition
* Not willing to have an X-ray
* Having blood vessels that are too difficult for inserting a cannula
* Having a hemoglobin of <8.4 mmol/L

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Concentrations of SCFAs | Between 0 and 10 hours
  (13C isotopic) enrichments of SCFAs inside intestinal lumen by GC-MS
Concentrations of plasma metabolites | Between 0 and 10 hours
  (13-C isotopic label incorporation) in plasma metabolites by GC-MS

SECONDARY OUTCOMES:
Concentrations of organic acids | Between 0 and 10 hours
  Organic acids measured in plasma and intestinal lumen by GC-MS
Concentrations of carbohydrates | Between 0 and 10 hours
  mono-, di-, tri-, oligo- and polysaccharides in the intestinal lumen by GC-MS
Concentrations of metabolites in urine | At baseline and after 10 hours
  bile acids, organic acids, amino acids by GC-MS
Concentrations of bile acids conjugates | Between 0 and 10 hours
Relative microbiota composition | Between 0 and 10 hours
  in the intestinal lumen, via 16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Guido Hooiveld, PhD, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Collected data will be coded

REFERENCES:
- [Background] den Besten G, Havinga R, Bleeker A, Rao S, Gerding A, van Eunen K, Groen AK, Reijngoud DJ, Bakker BM. The short-chain fatty acid uptake fluxes by mice on a guar gum supplemented diet associate with amelioration of major biomarkers of the metabolic syndrome. PLoS One. 2014 Sep 9;9(9):e107392. doi: 10.1371/journal.pone.0107392. eCollection 2014. PMID 25203112
- [Background] den Besten G, Lange K, Havinga R, van Dijk TH, Gerding A, van Eunen K, Muller M, Groen AK, Hooiveld GJ, Bakker BM, Reijngoud DJ. Gut-derived short-chain fatty acids are vividly assimilated into host carbohydrates and lipids. Am J Physiol Gastrointest Liver Physiol. 2013 Dec;305(12):G900-10. doi: 10.1152/ajpgi.00265.2013. Epub 2013 Oct 17. PMID 24136789